CLINICAL TRIAL: NCT05881564
Title: Differences in Outcomes for Patients (3.5-12kg) Undergoing Congenital Cardiac Surgery Who Receive Blood Versus Those Who do Not
Brief Title: Blood Conservation in Patients (3.5-12kg) Undergoing Congenital Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000190-3
Record Dates: First submitted 2023-05-10; First posted 2023-05-31 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Cardiopulmonary Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood prime for cardiopulmonary bypass (Active Comparator)
  Interventions: Other: blood use for priming cardiopulmonary bypass circuit
- clear prime for cardiopulmonary bypass (Active Comparator)
  Interventions: Other: clear prime for cardiopulmonary bypass

INTERVENTIONS:
Other: blood use for priming cardiopulmonary bypass circuit — one arm will have the cardiopulmonary bypass circuit primed with blood
  Arms: Blood prime for cardiopulmonary bypass
Other: clear prime for cardiopulmonary bypass — this arm will not have bypass circuit primed with blood
  Arms: clear prime for cardiopulmonary bypass

SUMMARY:
To evaluate if there is any clinical difference in patients 3.5-12kg who undergo cardiac surgery with cardiopulmonary bypass that do and do not receive blood products as part of their procedure. The main hypothesis of the study is that the patients undergoing bloodless cardiac surgery will have decreased morbidity and mortality when compared to the cohort that did receive blood as well as a shorter ICU and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Patient weight 3.5-12kg
* Elective and urgent cardiac surgery with cardiopulmonary bypass
* Cases within the STS STAT categories of 1-4

Exclusion Criteria:

* Patients who weigh more than 12kg or less than 3.5kg.
* Patients undergoing emergency surgery.
* STAT category 5 cases.
* Patients whose surgery does not require cardiopulmonary bypass.
* Patients presenting preoperatively in shock.
* Patients with known blood dyscrasias.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-05-11 (Estimated); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
Age of patients undergoing bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  age in months
Weight of patients undergoing bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  weight in kg
Gender of patients undergoing bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  sex
Demographics of bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  race
Diagnosis of patients undergoing bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  preoperative diagnosis
Surgery performed in bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  surgery performed
Previous surgery prior to bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  any previous surgery
Blood received during bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  blood product received
Volume transfused during bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  volume of blood transfusion in mL
Number of patients with unplanned reoperation in bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  unplanned reoperation
Number of patients with unplanned cardiac catheterization in bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  unplanned cardiac catheterization
Number of patients with a neurologic complication in bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  neurologic complication
Number of patients with chylothorax in bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  chylothorax
Number of patients with vocal cord injury in bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  vocal cord injury
Number of patients with diaphragm paralysis in bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  diaphragm paralysis
Number of patients with pacemaker implantation in bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  pacemaker implantation
Number of patients with postoperative pneumothorax in bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  postoperative pneumothorax
Number of patients with wound infection in bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  wound infection
Number of patients with bleeding requiring reoperation in bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  bleeding requiring reoperation
Number of patients with pericardial effusion in bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  pericardial effusion
Number of patients who died following bloodless cardiac surgery in patients 3.5-12kg (categorical variable) | 30 days
  mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Georgia, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No